CLINICAL TRIAL: NCT04400578
Title: TRICIN: Prospective Study on the Efficacy of Single Topical Trichloroacetic Acid (TCA) 85% in the Treatment of Cervical Intraepithelial Neoplasia (CIN 1/2)
Acronym: TRICIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Krankenhaus Barmherzige Schwestern Linz (Other)
Collaborators: Medical University of Vienna (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EKS 48/19
Record Dates: First submitted 2020-03-17; First posted 2020-05-22 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2020-03

CONDITIONS: Cervical Intraepithelial Neoplasia Grade 1; Cervical Intraepithelial Neoplasia Grade 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TRICIN (Experimental): If a patient is eligible
  1. local anesthesia with Xylocain 10% with a pump spray for a period of 10 seconds- one time application
  2. Procain 2%: local anesthesia with a swab for a period of 10 seconds- one time application
  3. Trichloroacetic acid TCA 85% 1-2 ml with soaked swab for max. 2 minutes -one time application
  Interventions: Device: Trichloroacetic acid 85% (TCA)

INTERVENTIONS:
Device: Trichloroacetic acid 85% (TCA) — Purpose and scope of Medical Device: Treatment and relief of a disease. Application to cervical intraepithelial neoplasia with a cotton swab.TCA is an investigational device intended to achieve a complete histologic remission in individuals with cervical intraepithelial neoplasia (CIN) grade 1/2.

SUMMARY:
Trichloroacetic acid 85% =TCA is an investigational device intended to achieve a complete histologic remission in individuals with cervical intraepithelial neoplasia (CIN) grade 1/2. The device system is to be used only in accordance with the approved Investigational Plan on subjects, who have given written informed consent.

High remission and regression rates are expected after a single topical treatment with 85% TCA. After a single topical treatment with 85% TCA for CIN 1-2 (Expected 70% or higher; null hypothesis: not higher than 55%). Regression is defined as improvement from high grade lesion (CIN 2) at baseline to low grade lesion (CIN 1) after TCA treatment. Regression from CIN 1 normal squamous epithelium after the TCA treatment is equal to remission and will be counted as a remission in combined analysis. Remission is defined as complete histologic remission of CIN back to normal squamous epithelium after the TCA treatment, i.e., no cervical dysplasia is detectable by histology or cytology after the TCA treatment. Type-specific HPV Clearance is defined as disappearance of the HPV type detected at screening.

DETAILED DESCRIPTION:
Visit and assessment Schedule:

Visit1 Screening:

* Informed Consent,
* Inclusion/Exclusion Criteria,
* Medical History,
* Gynecological Examination
* Cytology
* HPV Test
* Colposcopy
* Biopsy
* VAS (Visual analog scale)
* Pregnancy test

Visit 2 Treatment Day with TCA 85%:

* Colposcopy
* TCA Treatment
* VAS
* Pregnancy test

Visit 3, Control 1, Week 10-14:

* Cytology
* HPV Test
* Colposcopy
* Biopsy
* 4-quadrant biopsy
* ECC
* Adverse event monitoring If there is no sign of CIN during the colposcopic examination 10-14 weeks a 4-quadrant biopsy and a ECC are performed

Visit 4, Control 2, Week 22-26:

* Cytology
* HPV Test
* Colposcopy
* Biopsy
* 4-quadrant biopsy
* ECC
* Adverse event monitoring
* Pregnancy test If there is no sign of CIN during the colposcopic examination 22-26 weeks after the TCA treatment, a 4-quadrant biopsy and a ECC are performed.

Visit 5, EOS , Week 24-30:

- Results Discussion

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven CIN 1/2
* adequate colposcopy (i.e. fully visible transformation zone and margins of any visible lesion)
* positive HPV test
* conducted negative pregnancy test
* women aged 18 to 50 years
* written informed consent

Exclusion Criteria:

* Exclusion criteria are a cytologically suspected CIN (Pap IIID, IV)
* inadequate colposcopy
* negative or missing biopsy
* cytology results indicating invasive disease (PAP V)
* if the cervical lesion recedes into the endocervical canal
* pregnancy
* any medical circumstance considered relevant for proper performance of the study, or risks to the patient, at the discretion of the investigator

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 102 (Actual)
Dates: Start 2020-02-07 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2022-01-18 (Actual)

PRIMARY OUTCOMES:
CIN remission rate after treatment with TCA 85% | 6 months
  measured by histologic remission within 6 months

SECONDARY OUTCOMES:
CIN regression rate after treatment with TCA 85% | 6 months
  measured by histologic regression within 6 (improvement of at least one clinical CIN grade) months
Pain scores | 6 months
  measured by Visual Analogue Scale of a single use of TCA 85% in patients with CIN 1/2
Type specific human papillomavirus clearance rate after treatment with TCA 85% | 6 months
  human papillomavirus clearance rate after treatment with TCA 85% with CIN I/CIN // within 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Hefler, MD, Principal Investigator — Krankenhaus Barmherzige Schwestern Linz
Locations (1):
- Department of gynaecology, Ordensklinikum Linz Ges.m.b.H, Barmherzige Schwestern, Linz, Austria